CLINICAL TRIAL: NCT03400124
Title: Cost-effectiveness of Immediately Versus Delayed Sequential Bilateral Cataract Surgery (ISBCS vs. DSBCS)
Brief Title: Cost-effectiveness of ISBCS vs. DSBCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL64304.068.17
Record Dates: First submitted 2017-12-22; First posted 2018-01-17 (Actual); Last update posted 2021-09-05 (Actual); Status verified 2020-09

CONDITIONS: Bilateral Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ISBCS (Active Comparator): The intervention group will undergo cataract surgery of both eyes on the same day (ISBCS)
  Interventions: Procedure: ISBCS
- DSBCS (Active Comparator): The usual care / control group will undergo cataract surgery of both eyes on separate days, with a time period of at least two weeks between surgeries (DSBCS).
  Interventions: Procedure: DSBCS

INTERVENTIONS:
Procedure: ISBCS — The intervention group will undergo cataract surgery in both eyes on the same day (ISBCS)
  Arms: ISBCS
Procedure: DSBCS — The usual care / control group will undergo cataract surgery in both eyes on separate days, with a time period of at least two weeks between surgeries.
  Arms: DSBCS

SUMMARY:
The purpose of this study is to evaluate the effectiveness and costs of immediately sequential bilateral cataract surgery (ISBCS) compared to delayed sequential bilateral cataract surgery (DSBCS) in order to determine whether ISBCS is an effective and cost-effective alternative to DSBCS.

DETAILED DESCRIPTION:
With an estimated number of 180,000 cataract extractions per year in the Netherlands, cataract surgery is one of the most frequently performed types of surgery. The majority of patients suffer from bilateral cataract and while cataract surgery of one eye is effective in restoring functional vision, second-eye surgery leads to further improvement in health-related quality of life.

Currently, most patients undergo cataract surgery in both eyes on separate days as recommended in national guidelines, referred to as delayed sequential bilateral cataract surgery (DSBCS). An alternative procedure involves cataract surgery of both eyes on the same day, but as separate procedures, known as immediately sequential bilateral cataract surgery (ISBCS).

Potential benefits of ISBCS include less time between surgeries, a faster total recovery period and lower costs. Potential risks, however, are complications of cataract surgery in general, most importantly the risk of endophthalmitis and refractive surprise. In ISBCS, both eyes are at risk at the same time, while in DSBCS both eyes are exposed to these risks consecutively.

Since there is no consensus yet about the role of ISBCS in current regular practice, further investigation of functional and surgical outcomes and cost-effectiveness of ISBCS compared to DSBCS is required. Therefore, the purpose of this study is to evaluate the effectiveness and costs of ISBCS compared to DSBCS, in order to determine whether ISBCS is an effective and cost-effective alternative to DSBCS.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral cataract
* Indication for bilateral cataract surgery
* Expected uncomplicated surgery

Exclusion Criteria:

* Inability to comply with study procedures or to complete follow-up / Dutch questionnaires.
* Non-routine cataract surgery
* Cognitive or behavioural conditions that might interfere with surgery
* Cataract surgery with premium IOL implantation
* Conditions that increase the risk of endophthalmitis (e.g. current ocular/adnexal/periocular infections, immune-compromised, iodine allergy)
* Factors that increase the risk of refractive surprise (e.g. axial lengths <21mm or >27mm, difference between eyes of >1.5mm, abnormal keratometry readings, previous refractive surgery)
* Conditions that increase the risk of corneal edema
* Factors that increase the risk of complicated surgery (e.g. previous surgery, trauma, anatomical abnormalities)
* Sight-threatening comorbidity, Glaucoma or IOP > 24mmHg, Uveitis, Diabetes with diabetic retinopathy and macular edema

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 858 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Refraction: deviation of 1.0 D from target refraction | Four weeks post-operatively
  Proportion of patients in both treatment groups with a postoperative refraction in the second eye that deviates 1.0 diopters (D) from target refraction

SECONDARY OUTCOMES:
Refraction: deviation of 0.5 D from target refraction | Four weeks post-operatively
  Proportion of patients in both treatment groups with a postoperative refraction in the second eye that deviates 0.5 diopters (D) from target refraction
Change in visual acuity | Baseline, 1 week after first-eye surgery and 4 weeks after second-eye surgery
  Visual acuity will be measured by ETDRS letter charts
Complications | Intraoperatively and up to 4 weeks after second-eye surgery
  The incidence of intraoperative and postoperative complications
Patient reported outcome measures (PROMs): NEI VFQ-25 | Baseline and 3 months postoperatively
  Patient satisfaction and vision-specific quality of life as measured by National Eye Institute Visual Function Questionnaire (NEI VFQ-25).
Patient reported outcome measures (PROMs): Catquest | Baseline and 3 months postoperatively
  Patient satisfaction and vision-specific quality of life as measured by Catquest questionnaire.
Patient reported outcome measures (PROMs): HUI3 | Baseline, 1,4 weeks and 3 months postoperatively
  Health-related quality of life as measured by HUI3 (Health Utility Index Mark 3) questionnaire.
Patient reported outcome measures (PROMs): EQ-5D-5L | Baseline, 1,4 weeks and 3 months postoperatively
  Health-related quality of life as measured by EQ-5D-5L questionnaire.
Quality Adjusted Life Years (QALYs) | Baseline until 3 months postoperatively
  Calculated based on generic health-related quality of life, using the EQ-5D-5L and HUI-3 questionnaires
Costs per patient | Baseline until 3 months postoperatively
  Cost per patient, including valuation of resource use by using the Dutch guidelines for cost-analyses or cost prices provided by the medical center.
Incremental cost-effectiveness ratios (ICERs): QALY | Baseline until 3 months postoperatively
  Evaluation of cost-effectiveness by using calculated costs per quality-adjusted life years (QALYs)
Incremental cost-effectiveness ratios (ICERs): Target refraction | Baseline until 3 months postoperatively
  Calculated costs per patient with a postoperative refraction within 1.0 D of target refraction
Incremental cost-effectiveness ratios (ICERs): NEI VFQ-25 | Baseline until 3 months postoperatively
  Calculated costs per clinically improved patient on the NEI VFQ-25 questionnaire
Incremental cost-effectiveness ratios (ICERs): Catquest | Baseline until 3 months postoperatively
  Calculated costs per clinically improved patient on the Catquest questionnaire
Incremental cost-effectiveness ratios (ICERs): Visual acuity | Baseline until 3 months postoperatively
  Calculated costs per patient with clinical improvement in (un)corrected distance visual acuity
Budget impact | Baseline until 3 months postoperatively
  Reported as a difference in costs. Different scenario's will be compared to investigate the impact of various levels of implementation (e.g. 25%, 50%, 75% of eligible patients).

CONTACTS AND LOCATIONS:
Overall Officials: Rudy Nuijts, PhD, Principal Investigator — Department of Ophthalmology, Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center (MUMC+), Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Spekreijse L, Simons R, Winkens B, van den Biggelaar F, Dirksen C, Bartels M, de Crom R, Goslings O, Joosse M, Kasanardjo J, Lansink P, Ponsioen T, Reus N, Schouten J, Nuijts R. Safety, effectiveness, and cost-effectiveness of immediate versus delayed sequential bilateral cataract surgery in the Netherlands (BICAT-NL study): a multicentre, non-inferiority, randomised controlled trial. Lancet. 2023 Jun 10;401(10392):1951-1962. doi: 10.1016/S0140-6736(23)00525-1. Epub 2023 May 15. PMID 37201546
- [Derived] Spekreijse LS, Simons RWP, Winkens B, van den Biggelaar FJHM, Dirksen CD, Nuijts RMMA. Cost-effectiveness of immediate versus delayed sequential bilateral cataract surgery in the Netherlands (the BICAT-NL study): study design of a prospective multicenter randomised controlled trial. BMC Ophthalmol. 2020 Jun 29;20(1):257. doi: 10.1186/s12886-020-01521-x. PMID 32600295